CLINICAL TRIAL: NCT00873847
Title: Cerebral Function Monitoring and Brain Injury in Preterm Infants: Correlation With Neuroimaging Abnormalities and Neurodevelopmental Impairment - a Pilot Study
Brief Title: Cerebral Function Monitoring in Premature Infants
Status: Completed | Type: Observational
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: NICHD-NRN-0042; U10HD021373 (NIH); U10HD021385 (NIH); U10HD027851 (NIH); U10HD027880 (NIH); U10HD027904 (NIH); U10HD040492 (NIH); U10HD040689 (NIH); UL1RR025744 (NIH)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Electroencephalography
Keywords: NICHD Neonatal Research Network; Very Low Birth Weight (VLBW); Extremely Low Birth Weight (ELBW); Prematurity; Amplitude-integrated Electroencephalography (aEEG)
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This observational study tests the feasibility of enrolling subjects and obtaining an amplitude-integrated electroencephalogram (aEEG) within the first 72 hours of life, a second aEEG recording between 72-168 hours of life, and weekly thereafter up to 36 weeks post-menstrual age. It will enroll 85-100 infants between 401-1,000 grams birth weight OR between 23 0/7 and 28 6/7 weeks gestational age born at the 7 participating NICHD Neonatal Research Network sites.

DETAILED DESCRIPTION:
Few techniques exist to permit early and accurate prognosis of brain injury in newborns. Cranial ultrasound and magnetic resonance imaging (MRI) have been used to detect structural abnormalities which may be useful in predicting neuromotor and neurocognitive deficits. However, up to 30% of extremely low birth weight infants with normal ultrasounds have adverse outcomes, and MRI is not feasible when an infant is critically ill. Amplitude-integrated electroencephalogram (aEEG) is a non-invasive, bedside instrument which allows real-time monitoring of brain function and may provide additional information for predicting outcomes in extremely premature infants.

This observational study will enroll 85-100 infants between 401-1,000 grams birth weight OR between 23 0/7 and 28 6/7 weeks gestational age born at the 7 participating NICHD Neonatal Research Network sites. Eligible infants will undergo an aEEG recording in the first 72 hours of life, a second aEEG recording between 72-168 hours of life, and weekly thereafter up to 36 weeks post-menstrual age.

The study tests the feasibility of enrolling subjects and obtaining the required aEEG recordings. The information gathered will provide a framework for the design of a potential prospective, observational, multi-center study for prediction of death or neurodevelopmental impairment by 18-22 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Inborn infants
* Between 401 grams and 1,000 grams inclusive birth weight OR between 23 0/7 and 28 6/7 weeks inclusive gestational age
* Decision to provide full intensive care support
* Less than 72 hours of age

Exclusion Criteria:

* Non-intact skin at the central or parietal regions of scalp
* Presence of known or suspected congenital anomalies, including:
* Congenital central nervous system malformations
* Chromosomal anomalies or multiple congenital anomalies
* Complex congenital heart disease
* Inborn error of metabolism
* Acidosis (pH < 6.8 for > 2 hours)
* Persistent bradycardia [HR < 100 bpm] associated with hypoxia for > 2 hours

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants born at NRN centers and admitted to the NICU that are between 401 grams and 1,000 grams OR between 23 0/7 and 28 6/7 weeks gestational age. Infants must be enrolled by the time they are 72 hours old.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
First aEEG within 72 hours of age | < 72 hours of age

SECONDARY OUTCOMES:
Time required by research personnel to conduct study activities | Birth to 36 weeks post menstrual age
Serious adverse events | < 72 hours of age until 36 weeks post menstrual age
Agreement between aEEG recordings and clinical events including: seizures, cardiopulmonary resuscitation, surfactant administration, suctioning, and intubation | < 72 hours of age until 36 weeks post menstrual age
Weekly aEEG until infant is 36 weeks post menstrual age | < 72 hours of age until 36 weeks post menstrual age

CONTACTS AND LOCATIONS:
Overall Officials: Abbot R. Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Ricki F. Goldstein, MD, Principal Investigator — Duke University; Barbara J. Stoll, MD, Principal Investigator — Emory University; Abhik Das, PhD, Principal Investigator — RTI International; Alexis Davis, MD, Principal Investigator — Stanford University; Lina Chalak, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Kathleen A. Kennedy, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Seetha Shankaran, MD, Principal Investigator — Wayne State University
Locations (8):
- United States (8):
  - Stanford University, Palo Alto, California
  - Emory University, Atlanta, Georgia
  - Wayne State University, Detroit, Michigan
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas

REFERENCES:
- [Result] Davis AS, Gantz MG, Do B, Shankaran S, Hamrick SE, Kennedy KA, Tyson JE, Chalak LF, Laptook AR, Goldstein RF, Hintz SR, Das A, Higgins RD, Ball MB, Hale EC, Van Meurs KP; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Serial aEEG recordings in a cohort of extremely preterm infants: feasibility and safety. J Perinatol. 2015 May;35(5):373-8. doi: 10.1038/jp.2014.217. Epub 2014 Dec 4. PMID 25474559
- See also: NICHD Neonatal Research Network — https://neonatal.rti.org/